CLINICAL TRIAL: NCT03042000
Title: A Multicenter, Prospective, Randomized Clinical Trial to Investigate the Combined Modality Therapy for Locally Advanced Mid/Low Rectal Cancer.
Brief Title: Multicenter, Prospective, RCT：Investigation of Combined Modality Therapy for Locally Advanced Mid/Low Rectal Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Chao Yang Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Beijing Friendship Hospital (Other); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Guole Lin, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-Colorectal Surgery 02
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Rectal Cancer, Adenocarcinoma; Neoadjuvant Chemoradiation
Keywords: rectal cancer; neoadjuvant chemoradiation; circulating tumor DNA; local recurrence; long-term survival
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A1 (Experimental): Patients with cT3a-bN0-1aM0 mid rectal cancer who undergo the treatment modality of 'radical surgery + adjuvant chemotherapy (ACT)'
  Interventions: Other: non-NCRT
- Group A2 (Active Comparator): Patients with cT3a-bN0-1aM0 mid rectal cancer who undergo the treatment modality of 'NCRT + radical surgery + ACT'
  Interventions: Other: NCRT
- Group B1 (Experimental): Patients with cT4NanyM0 or cTanyN2M0 mid/low rectal cancer who undergo the treatment modality of 'NCRT with combined chemotherapy (Capox regimen) + radical surgery + ACT'
  Interventions: Drug: capecitabine with oxaliplatin
- Group B2 (Active Comparator): Patients with cT4NanyM0 or cTanyN2M0 mid/low rectal cancer who undergo the treatment modality of 'NCRT with single-agent chemotherapy (Capecitabine) + radical surgery + ACT'
  Interventions: Drug: capecitabine
- Group C1 (Experimental): Patients with locally advanced rectal cancer, being clinically staged cCR after NCRT, who undergo the transanal endoscopic microsurgery (TEM) excision of the lesion.
  Interventions: Procedure: TEM
- Group C2 (Active Comparator): Patients with locally advanced rectal cancer, being clinically staged cCR after NCRT, who undergo the radical resection of the lesion.
  Interventions: Procedure: radical resection

INTERVENTIONS:
Other: non-NCRT — without the preoperative concurrent chemoradiothearpy (no neoadjuvant chemoradiation)
  Arms: Group A1
Other: NCRT — the preoperative concurrent chemoradiothearpy (neoadjuvant chemoradiation)
  Arms: Group A2
Drug: capecitabine with oxaliplatin — combined chemotherapy with capecitabine with oxaliplatin
  Arms: Group B1
Drug: capecitabine — single-agent chemotherapy with capecitabine
  Arms: Group B2
Procedure: TEM — transanal endoscopic microsurgery (TEM) excision of the lesion
  Arms: Group C1
Procedure: radical resection — radical resection of rectal cancer
  Arms: Group C2

SUMMARY:
At present, the combined modality treatment of preoperative neoadjuvant chemoradiotherapy (NCRT) followed by radical surgery has become the standard of care for the locally advanced mid/low rectal cancer, having been proved to substantially improve the local control of the disease, whereas not being able to improve the long-term survival. According to present clinical practice guidelines, all patients with cT3-4N0M0 or cTanyN1-2M0 mid/low rectal cancer are recommended to undergo the preoperative long-term radiotherapy with concurrent 5FU based chemotherapy, followed by the radical resection of the tumor. After surgery, adjuvant chemotherapy (ACT) is recommended for all these patients without considering the postoperative pathological results. Recently, however, some authors proposed that different strategy of combined modality therapy should be applied in different patients according to their risk of relapse, instead of using the uniform NCRT strategy. In this research, on the basis of investigator's previous clinical practice and researches, investigators plan to stratify the patients with cT3-4N0M0 or cTanyN1-2M0 mid/low rectal cancer into several subgroups according to tumor stages and the risk of relapse. Different therapeutic strategy will be applied in different groups, at the aim of improving the overall therapeutic effects, as well as reducing the treatment adverse effects.

This research consists of four trials.

DETAILED DESCRIPTION:
Trial A: A multicenter, prospective, randomized trial to compare neoadjuvant chemoradiotherapy (NCRT) followed by radical surgery with surgery alone for cT3a-bN0-1aM0 mid rectal cancer.

Research objects: Patients with locally advanced rectal cancer, being clinically staged T3a-bN0-1aM0 by rectal MRI and/or endorectal ultrasonography (ERUS), the tumor being located 6-12 cm above the anal verge.

After giving fully informed consent, the prospective participants will be randomly divided into two groups, receiving the following two treatment modalities.

Group A1: radical surgery + adjuvant chemotherapy (ACT) Group A2: NCRT + radical surgery + ACT

Trial B: A multicenter, prospective, randomized trial to compare combined versus single-agent chemotherapy with concurrent radiotherapy for cT4NanyM0 or cTanyN2M0 rectal cancer.

Research objects: Patients with locally advanced rectal cancer, being clinically staged cT4NanyM0 or cTanyN2M0 by rectal MRI and/or ERUS, or patients with any other risk factors for tumor relapse.

After giving fully informed consent, the prospective participants will be randomly divided into two groups, receiving the following two treatment modalities.

Group A1: NCRT with combined chemotherapy (Capox regimen) + radical surgery + ACT Group A2: NCRT with single-agent chemotherapy (Capecitabine) + radical surgery + ACT

Trial C: A multicenter, prospective, randomized trial to compare transanal ndoscopic microsurgery (TEM) excision versus radical resection of rectal cancer being staged clinical complete response (cCR) after NCRT.

Research objects: Patients with locally advanced rectal cancer, being clinically staged cCR after NCRT.

After giving fully informed consent, the prospective participants will be randomly divided into two groups, receiving the following two treatment modalities.

Group A1: TEM excision + ACT Group A2: radical surgery + ACT

Trial D: A prospective, observational study to determine the value of circulating tumor DNA (ctDNA) for predicting the therapeutic effects of NCRT for locally advanced rectal cancer and the patients' long-term prognosis.

Research objects: Patients with locally advanced mid/low rectal cancer (cT3-4N0M0 or cTanyN+M0) who undergo NCRT.

After giving fully informed consent, the prospective participants will undergo the classical 'NCRT + radical surgery + ACT' comprehensive treatment. Serial analysis of ctDNA will be performed at specific time points including pre-NCRT, post-NCRT, postoperative week 1, post-ACT, postoperative year 1, 2, and 3. The next-generation sequencing of surgical specimens will be performed as well. Participants will be observed and examined during the entire course of treatment and the follow-up period. The pathological results of the surgical specimen and the 3 year disease free survival (3y-DFS) will be the main end-points.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 75 years old. Patients with cT3-4N0M0 or cTanyN+M0 mid/low rectal cancer. Patients with ASA physical status scroe of I to III. Patients who can fully understand the content of the informed consent form and sign it upon their own opinions.

Patients who can coordinate with the researchers to undergo the long-term post-treatment rechecks and follow-ups.

Exclusion Criteria:

Patient has any underlying or current medical condition, which, in the opinion of the Investigator, would interfere with the evaluation of the patient (e.g., end-stage liver disease, pulmonary hypertension, systemic lupus erythematosis etc.).

Patient is pregnant or lactating. Patient has a history of malignancy within 5 years except curatively treated basal cell carcinoma, squamous cell carcinoma in a non-mucosal, ultraviolet exposed area, or cervical carcinoma.

Patient is participating in any other clinical trials within 30 days prior to screening.

Patient has severe mental illness. Patient has any other conditions, which, in the opinion of the Investigator, would interfere with the evaluation of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
3y-DFS | 3 years
  the 3-year disease free survival rate

SECONDARY OUTCOMES:
3y-OS | 3 years
  the 3-year overall survival rate
5y-DFS | 5 years
  the 5-year disease free survival rate
5y-OS | 5 years
  the 5-year overall survival rate
pCR | 4 months
  pathological complete tumor response rate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou J, Qiu H, Lin G, Xiao Y, Wu B, Wu W, Sun X, Lu J, Zhang G, Xu L, Liu Y. Is adjuvant chemotherapy necessary for patients with pathological complete response after neoadjuvant chemoradiotherapy and radical surgery in locally advanced rectal cancer? Long-term analysis of 40 ypCR patients at a single center. Int J Colorectal Dis. 2016 Jun;31(6):1163-8. doi: 10.1007/s00384-016-2579-5. Epub 2016 Apr 5. PMID 27044403
- [Background] Ferrari L, Fichera A. Neoadjuvant chemoradiation therapy and pathological complete response in rectal cancer. Gastroenterol Rep (Oxf). 2015 Nov;3(4):277-88. doi: 10.1093/gastro/gov039. Epub 2015 Aug 19. PMID 26290512
- [Background] Breugom AJ, Swets M, Bosset JF, Collette L, Sainato A, Cionini L, Glynne-Jones R, Counsell N, Bastiaannet E, van den Broek CB, Liefers GJ, Putter H, van de Velde CJ. Adjuvant chemotherapy after preoperative (chemo)radiotherapy and surgery for patients with rectal cancer: a systematic review and meta-analysis of individual patient data. Lancet Oncol. 2015 Feb;16(2):200-7. doi: 10.1016/S1470-2045(14)71199-4. Epub 2015 Jan 12. PMID 25589192
- [Background] Bosset JF, Calais G, Mineur L, Maingon P, Stojanovic-Rundic S, Bensadoun RJ, Bardet E, Beny A, Ollier JC, Bolla M, Marchal D, Van Laethem JL, Klein V, Giralt J, Clavere P, Glanzmann C, Cellier P, Collette L; EORTC Radiation Oncology Group. Fluorouracil-based adjuvant chemotherapy after preoperative chemoradiotherapy in rectal cancer: long-term results of the EORTC 22921 randomised study. Lancet Oncol. 2014 Feb;15(2):184-90. doi: 10.1016/S1470-2045(13)70599-0. Epub 2014 Jan 17. PMID 24440473
- [Background] Vogelstein B, Papadopoulos N, Velculescu VE, Zhou S, Diaz LA Jr, Kinzler KW. Cancer genome landscapes. Science. 2013 Mar 29;339(6127):1546-58. doi: 10.1126/science.1235122. PMID 23539594
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Zhou J, Chang L, Guan Y, Yang L, Xia X, Cui L, Yi X, Lin G. Application of Circulating Tumor DNA as a Non-Invasive Tool for Monitoring the Progression of Colorectal Cancer. PLoS One. 2016 Jul 26;11(7):e0159708. doi: 10.1371/journal.pone.0159708. eCollection 2016. PMID 27459628
- [Background] Reinert T, Scholer LV, Thomsen R, Tobiasen H, Vang S, Nordentoft I, Lamy P, Kannerup AS, Mortensen FV, Stribolt K, Hamilton-Dutoit S, Nielsen HJ, Laurberg S, Pallisgaard N, Pedersen JS, Orntoft TF, Andersen CL. Analysis of circulating tumour DNA to monitor disease burden following colorectal cancer surgery. Gut. 2016 Apr;65(4):625-34. doi: 10.1136/gutjnl-2014-308859. Epub 2015 Feb 4. PMID 25654990
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Jung KU, Kim HC, Park JO, Park YS, Park HC, Choi DH, Cho YB, Yun SH, Lee WY, Chun HK. Adjuvant chemotherapy after neoadjuvant chemoradiation and curative resection for rectal cancer: is it necessary for all patients? J Surg Oncol. 2015 Mar 15;111(4):439-44. doi: 10.1002/jso.23835. Epub 2014 Dec 9. PMID 25488390